CLINICAL TRIAL: NCT04062747
Title: Comparison Of The Effect Of I-Gel And Ambu Aura-I Use On Laryngofaryngeal Mucosa Wıth Flexible Bronchoscopy in Infants
Brief Title: The Effect Of I-Gel And Ambu Aura-I Use On Laryngofaryngeal Mucosa
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 71306642-S001
Record Dates: First submitted 2019-08-08; First posted 2019-08-20 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Mucosal Damage
Keywords: Laryngeal Mask; I-gel; Ambu Aura i; Flexible bronchoscopy; Laryngopharyngeal damage; Infant

STUDY DESIGN:
Intervention Model Description: Mucosal damage and postoperative complications in laryngopharyngeal structures were compared.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- I-gel LMA (Active Comparator): After standard anesthesia i-Gel was placed into the patient.
  Interventions: Device: I-gel
- Ambu Aura-i (Active Comparator): After standard anesthesia Ambu Aura-i was placed into the patient.
  Interventions: Device: Ambu aura i

INTERVENTIONS:
Device: I-gel — After standard anesthesia i-Gel was placed into the patient
  Other Names: I-gel laryngeal mask airway
  Arms: I-gel LMA
Device: Ambu aura i — After standard anesthesia ambu aura was placed into the patient
  Other Names: Ambu aura i laryngeal mask airway
  Arms: Ambu Aura-i

SUMMARY:
Supraglottic airway devices (SGADs) are frequently preferred in surgical surgery for pediatric patients. i-gel LMA (laryngeal mask airway) and Ambu Aura-i LMA are the new generation supraglottic airway devices. The aim of this study was to compare airway trauma and postoperative complications due to i-gel and Ambu Aura in infants. In the study patients were divided into two groups performed on minor surgery ASA I (American Society of Anesthesiologists score) and 40 infants. After standard anesthesia i-Gel was placed into a group and Ambu Aura-i was placed to the other. Flexible bronchoscopy was performed at the end of surgery. Mucosal damage and postoperative complications in laryngopharyngeal structures were compared.

DETAILED DESCRIPTION:
This study was conducted as prospective, randomized and double-blind study. After confirmation the approval from the Interventional Ethics Committee of the Bezmialem Vakif University, dated…. Number…., the study was started. Forty ASA I patients under the age of 1, with a body weight of more than 10 kg, without anatomical pathology in the upper airway with no general anesthesia within the last 2 weeks who underwent minor surgery (circumcision, inguinal hernia, undescended testis, hypospadias, etc.) by the Pediatric Surgery Clinic at Bezmialem Vakif University Medical School Hospital were included in the study. Patients who are older than 1 year of age and have a body weight of more than 10 kg, who have symptoms of upper or lower respiratory tract infection, who have more than one trial performed during the SADs placement, who are known and expected to be difficult airway, who has undergone surgery for more than 2 hours and patients who underwent emergency surgery were not included in the study.

ELIGIBILITY:
Inclusion Criteria:

1. ASA I
2. patients under the age of 1,
3. body weight of less than 10 kg
4. without anatomical pathology in the upper airway
5. no general anesthesia within the last 2 weeks who underwent minor surgery

Exclusion Criteria:

1. older than 1 year of age
2. body weight of more than 10 kg
3. symptoms of upper or lower respiratory tract infection
4. more than one trial performed during the SADs placement
5. known and expected to be difficult airway
6. undergone surgery for more than 2 hours and patients
7. underwent emergency surgery

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2019-05-18 (Actual); Primary Completion 2019-09-15 (Estimated); Study Completion 2019-09-20 (Estimated)

PRIMARY OUTCOMES:
airway trauma | up to 1 minute after extubation
  4 point scoring system 1- no hyperemia 2- mild hyperemia 3- severe hyperemia 4-mucosal damage and bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakıf University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No